CLINICAL TRIAL: NCT05884177
Title: Metabolic Effects of Short-term Cold Exposure Among Greenlanders and Non-Greenlanders
Brief Title: Inuit and Cold Exposure
Acronym: ICE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Stig Andersen (Other)
Collaborators: University of Copenhagen (Other); Greenland University (Unknown)
Responsible Party: Sponsor-Investigator, Stig Andersen, Professor, Department Head, Aalborg University Hospital
Organization: Aalborg University Hospital (Other)
Other Study IDs: F2023-040
Record Dates: First submitted 2023-05-04; First posted 2023-06-01 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Healthy
Keywords: Brown Adipose Tissue

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Greenlanders: Subjects born in Greenland with parents born in Greenland
  Interventions: Other: Short-term cold exposure
- non-Greenlanders: Subjects not born in Greenland with parents not born in Greenland
  Interventions: Other: Short-term cold exposure

INTERVENTIONS:
Other: Short-term cold exposure — Short-term cold exposure

SUMMARY:
Brown adipose tissue (BAT) produces heat through non-shivering thermogenesis. It is activated by cold exposure, and when activated it utilizes fatty acids and glucose in order to produce heat. The tissue is especially present in newborns, who not yet have gained a layer of insulating fat to protect from heat loss, and not yet have gained much muscle to produce heat through shivering thermogenesis.

It was long thought that BAT mass hereafter would retract. Modern imaging tools have proved that BAT is persistent and active in some adults. The presence and activity of BAT is negatively correlated with obesity and obesity-related metabolic disorders. The tissue retracts with advancing age and increasing BMI, and it is sensitive to environmental factors, such as diet, weather and climate. The key to activating BAT in subjects that have lost it remains elusive.

BAT is activated to produce heat when exposed to cold. Populations that are most cold exposed include people living in the Arctic. It is known that people of Arctic origin such as indigenous Inuit and indigenous Siberians have genetically adapted to and are acclimatized to the cold through several genetic changes, and possibly by upregulating BAT depots and activity. The investigators aim to dig deeper into the activation mechanisms in BAT, by investigating BAT mass and activity in Greenlanders and non-Greenlanders by use of stage-of-the-art modern techniques.

DETAILED DESCRIPTION:
Several studies have examined the function of brown adipose tissue (BAT), which is an important source of non-shivering thermogenesis. It has gained attention as a potential target for combating obesity.

BAT has a distinct influence on glucose and triglyceride clearance, and insulin sensitivity, and it has a negative correlation with cardiometabolic risk markers.

BAT activity is correlated with cold temperatures. Observational studies in Greenland are consistent with raised consumption of thyroid hormone and higher thyroid hormone turnover in cold-exposed Inuit compared to Inuit with some and limited cold exposure.

However, these are indirect data that merely suggest the presence of BAT. The presence of active BAT directly illustrated by using an individualized cooling protocol and FDG-PET/CT-scan raises interest in the origin and characterization of intermediate adipose cells (beige adipose tissue) from the white adipose tissue.

Based on the strong correlation between BAT and cardiometabolic health and the evolutionary pressure on Inuit to handle cold environments, the investigators will measure the cold-induced BAT activity and white fat differentiation and assess a connection with genetic and physiological characteristics ot add insight into the biology and regulation of BAT in relation to fat depots in humans.

Participants of Danish and Greenlandic origin will be included for a focus on visualizing brown adipose tissue by use of PET/CT-scans before and after short term cold exposure. Additional sampling includes subcutaneous fat biopsies, blood samples, blood pressure, pulse, temperature of the skin and core, and IRT.

ELIGIBILITY:
Inclusion Criteria:

* Ability to give informed consent
* Ability to follow written and verbal instructions

Exclusion Criteria:

* Pregnancy and breastfeeding
* Alpha- or beta-adrenergic affecting medication.
* Thyroid dysfunction
* Liver or kidney disease
* Treatment for diabetes
* MODY and TBC1D4
* Treatment of obesity
* Cardiovascular disease
* Cancer within 3 years
* Mb Renaud
* Hospitalisation for psychiatric disease
* Antipsychotic medication
* Drug abuse within 1-year
* Alcohol abuse
* Plasma glucose > 11 mM
* BMI >35 kg/m2
* Winter swimmer

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy, lean, young Greenlanders and non-Greenlanders living in Denmark
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2023-09-18 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
BAT detection | Through study completion, analysis for an average of 1 year
  BAT mass in the cervical-upper thoracic, abdominal, and paravertebral regions at room temperature and following short-term cold exposure. BAT mass on PET/CT scans will be quantified by the degree of glucose uptake: Maximum standard unit value (SUVmax)

SECONDARY OUTCOMES:
Temperature of the core and at the skin on multiple sites | Through study completion, analysis for an average of 1 year
  Temperature of the core and at the skin on multiple sites. Core temperature measured with rectal thermometer. Skin temperatures measured with skin thermometer probes and infrared thermography (IRT).
Changes in thyroid function | Through study completion, analysis for an average of 1 year
  Changes in thyroid function as measured by plasma TT3, TT4 and TSH
Changes in metabolites | Through study completion, analysis for an average of 1 year
  Changes in metabolites: Plasma glucose, acylcarnitine and triglycerides
Insulin sensitivity | Through study completion, analysis for an average of 1 year
  Insulin sensitivity
Adipose tissue composition | Through study completion, analysis for an average of 1 year
  Subcutaneous fat biopsies will be examined in relation to white adipose tissue (WAT) function and presence of beige adipocytes

CONTACTS AND LOCATIONS:
Locations (1):
- Aalborg University Hospital, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No
Restrictions apply due to limited number of participants

REFERENCES:
- [Derived] Motzfeldt Jensen M, Almasi CE, Kjaergaard B, Rasmussen BS, Andersen MK, Schubert M, Hansen T, Ellervik C, Scheele C, Jorgensen ME, Andersen S. Brown Adipose Tissue and Metabolic Markers Differ Between Greenlanders and Danes with Cold-Activation. J Clin Endocrinol Metab. 2025 Nov 17:dgaf615. doi: 10.1210/clinem/dgaf615. Online ahead of print. PMID 41243523